CLINICAL TRIAL: NCT04489095
Title: Evaluation of Conduction Disease After Trans-catheter Aortic Valve Replacement
Brief Title: Conduction Disease After Transcatheter Aortic Valve Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Tiberio Frisoli, MD Principal Investigator, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Frisoli_13944
Record Dates: First submitted 2020-05-28; First posted 2020-07-28 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Aortic Stenosis; Heart Block; Aortic Insufficiency
Keywords: Transcatheter Aortic Valve Replacement; TAVR; Aortic stenosis; AS; Pacemaker; HV interval; Electrophysiology Study; EPS; Heart block
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Block; Aortic Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: After informed consent is obtained, patient will undergo TAVR as per usual standard of care. Using the same femoral vein access as is used standard for a portion of the TAVR procedure, an EPS(Electrophysiology study) will be performed during the TAVR procedure, immediately before and after valve implantation. The patient will recover on a general telemetry floor as per usual care, and the next day will undergo another EPS. This is not uncommonly done clinically for some patients after TAVR. At that point, based on the baseline EKG, intra-procedure findings, and EPS findings, the patient will either have a pacemaker implanted, a 30-day event monitor ordered, or neither of the above.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Electrophysiology Study pre and Post TAVR (Experimental): In all patient's undergoing TAVR after informed consent will undergo an electrophysiology study pre and post device deployment in order to determine the need for permanent pacemaker implantation or further testing/monitoring.
  Interventions: Diagnostic Test: Electrophysiology Study

INTERVENTIONS:
Diagnostic Test: Electrophysiology Study — After informed consent is obtained, patient will undergo TAVR as per usual standard of care. Using the same femoral vein access as is used standard for a portion of the TAVR procedure, an EPS will be performed during the TAVR procedure, immediately before and after valve implantation. The patient will recover on a general telemetry floor as per usual care, and the next day will undergo another EPS. This is not uncommonly done clinically for some patients after TAVR. At that point, based on the baseline EKG, intra-procedure findings, and EPS findings, the patient will either have a pacemaker implanted, a 30-day event monitor ordered, or neither of the above.

SUMMARY:
This is a prospective single center Cardiology department observational study. The study aim is to better understand the predictors of high grade conduction abnormalities associated with TAVR such that a more robust evidence-based and universal strategy to manage cardiac conduction disturbances in these patients, which has been elusive, can be developed.

DETAILED DESCRIPTION:
TAVR is a very commonly performed procedure throughout the world; it has become standard of care as the treatment for aortic stenosis and is performed in hundreds of thousands of patients annually. TAVR affords patients therapies that prolong life and improve quality of life; furthermore, these therapies afford certain patients who are not candidates for surgical options hope for the future. Adults undergoing TAVR may suffer the complication of requiring a pacemaker after the procedure, in up to 30% of cases. Interventionalists still don't understand how to best predict this complication; in fact some patients that ultimately need a pacemaker don't get one after the procedure and some that get a pacemaker are found to ultimately not have really needed it. A better understanding of which patients do and do not need pacemakers will help prevent complications of high grade block in those without pacemaker (death, syncope and trauma) and also the complications of unnecessary pacemaker implantation (infection, tricuspid regurgitation).

Primary hypothesis: EP studies (EPS), when performed before and after TAVR adds independent incremental value, above and beyond other parameters, for the prediction of high-grade heart block after TAVR. The goal is to understand conduction disease changes before and after TAVR, coupled with other patient and procedural factors that can help create a management algorithm for conduction disease after TAVR.

Primary endpoint: to find correlation coefficients between a) absolute and delta values of various EPS findings, and b) clinical endpoint of high-grade conduction disease as diagnosed clinically, by ECG, by event monitor, or by interrogation of permanent pacemaker implanted after TAVR.

Methods: Patients will receive EPS immediately before and after TAVR (while on the catheterization lab table for TAVR procedure) and then again the next day; this information will help determine whether the patient gets a pacemaker, a 30-day event monitor, or neither. The investigators will study which parameters obtained during the EPS, in addition to other known/suspected predictors of conduction disease after TAVR, best correlate with serious problems with the heart's electrical conduction system as determined by clinical follow-up.

Anticipated findings: that the EPS findings add incremental and independent value in predicting which patients will develop high grade conduction disease.

ELIGIBILITY:
Inclusion Criteria

* Signed and dated Informed Consent
* Patient that undergoes a TAVR
* Ability to complete functional assessments.

Exclusion Criteria:

* Patients with pre-existing permanent pacemaker.
* Patient unwilling or unable to follow-up for necessary pre- and post-procedure clinical assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
High grade conduction disease post TAVR | 1 year
  Number of participants that develop high grade conduction block post TAVR including complete heart block, 2nd degree AV block, symptomatic bradycardia

SECONDARY OUTCOMES:
death | 1 year
  Rate of mortality by chart review and SSDI query at 1 year
rehospitalization | 1 year
  Absolute and per patient hospitalizations post index procedure
need for pacemaker implantation | 1 year
  Percentage of participants requiring permanent pacemaker implantation in index hospitalization or within 1 year
HV interval pre and post TAVR | 2 days
  Absolute HV interval in milliseconds as measure by electrophysiology study for each participant pre and post TAVR
ejection fraction | 1 year
  Ejection fraction as measured by trans-thoracic echocardiography for each participant pre and post tavr on routine trans-thoracic echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Tiberio Frisoli, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No